CLINICAL TRIAL: NCT03794076
Title: Cromoglicte Adjunctive Therapy for Outpatients With Schizophrenia
Brief Title: Cromoglicate Adjunctive Therapy for Outpatients With Schizophrenia
Acronym: CATOS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vishwajit Nimgaonkar, MD PhD (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19070355
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Schizo Affective Disorder
Keywords: schizophrenia; schizoaffective disorder; cromoglicate
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cromolyn Sodium

STUDY DESIGN:
Intervention Model Description: This study will be a randomized placebo-controlled sequential parallel comparison design (SPCD).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care providers, Investigators and assessors will all be blinded. Study staff responsible for randomization will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cromoglycate (Active Comparator): Cromoglycate nasal spray
  Interventions: Drug: Cromoglycate; Drug: Placebo
- Placebo (Placebo Comparator): Saline nasal spray
  Interventions: Drug: Cromoglycate; Drug: Placebo

INTERVENTIONS:
Drug: Cromoglycate — Cromoglycate will be administered intranasally (nasal spray) (1 spray each nostril 4 times a day, 5.2 mg/spray
  Other Names: NasalCrom
Drug: Placebo — Normal saline nasal spray will be administered intranasally (nasal spray) (1 spray each nostril 4 times a day, 5.2 mg/spray)
  Other Names: Saline Nasal Spray

SUMMARY:
This is a double blind adjunctive randomized controlled trial for schizophrenia using cromoglicate.

DETAILED DESCRIPTION:
Schizophrenia (SZ) extracts a heavy personal and public health cost, primarily because there is no effective treatment. Though many drugs are currently available, the majority provide only partial relief for psychotic phenomena and none guarantee more than modest relief for 'negative symptoms' or for cognitive impairments. The Investigators must search for additional effective and safe medications. Recently, big data analytic strategies have yielded numerous 'repurposed' drugs, i.e., drugs with new indications that are already licensed for other uses. These strategies utilize massive data bases of known drug effects to find candidates that could predictably counteract known pathogenic effects of the disorder in question. Repurposed drugs are appealing not only because they have already been marketed and have known side effect profiles, but also because they have increased prior probability of efficacy. Still, careful randomized controlled trials (RCTs) are necessary for the new indications. The investigators have designed a systematic search for repurposed drugs likely to be beneficial for patients with SZ. Our novel search strategy began with the construction of a comprehensive protein-protein interaction network (PPI) for SZ using a validated method. Next, The Investigators searched public data bases for drugs that have predicted effects on multiple proteins in the SZ PPI network, but opposite to those observed in patients with SZ. The initial list was pruned using predetermined criteria, leaving 7 drugs of which cromoglycate (CGY) had the best negative correlation score. Reassuringly, three other drugs with lower scores in our list have already been tested for SZ. CGY is a safe and highly effective mast cell inhibitor that has been licensed for over 25 years for prophylaxis of asthma and allergies; it is also used to treat systemic mastocytosis and ulcerative colitis. Independent of our research, CGY is also predicted to stabilize the blood brain barrier (BBB), which can be disrupted in patients with SZ. Animal studies and favorable Log P estimates assure that CGY can cross the BBB. CGY has few reported side effects, despite its extensive use. Thus, multiple factors motivate our RCT. The Investigators propose a double blind adjunctive RCT for SZ using CGY. To maximize therapeutic benefits while minimizing risk and discomfort, The Investigators will enroll outpatients with SZ who meet criteria for residual positive symptoms after adequate trials of standard antipsychotic drug (APD) therapy (N=100, total). The Investigators will prefer patients in the early course of their illness. CGY or placebo will be added to prescribed medications for 4 weeks utilizing the Sequential Parallel Comparison Design to maximize power. The primary outcome will be improvement in positive symptoms as determined by the Positive and Negative Syndrome Scale (PANSS) positive symptom subscale. Secondary outcomes include total symptoms (PANSS total score), negative symptoms (PANSS negative symptom scale scores), cognition (Penn Computerized Neurocognitive Battery), and social function. Serum CGY levels will be monitored. The Investigators have proven experience with RCTs and the large number of patients are our clinical service ensures that recruitment targets will be fulfilled.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Both genders, ages 18-60 years
* Schizophrenia / schizoaffective disorder (DSM V).
* Treated with the same APD for at least 60 days; Stable dose of APD for > 1 month, continued throughout the study.
* PANSS total score of 60 and Score 4 or more on one or more items of the 'positive' syndrome items (P1-P7)
* Preference for patients with duration of psychosis less than 7 years.

Exclusion Criteria:

* No illicit substance use in last 30 days/no dependence in 6 months with the exception of methadone treatment for opioid withdrawal.
* History or current medical /neurological illnesses that may lead to an unstable course with the exception of epilepsy which is well-controlled on an antiepileptic medication for at least 6 months.
* Pregnancy.
* History of immune disorders, HIV infection, or receiving immune-suppressants or immuno-modulators, e.g., steroids.
* Current or prior treatment with CGY or History of hypersensitivity to CGY.
* Intellectual disability as defined in DSM V.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in positive symptoms | 12 weeks
  Clinical Severity as determined by the Positive and Negative Syndrome Scale (PANSS) positive symptom subscale. The PANSS is a standardized, clinical interview that rates the presence and severity of positive and negative symptoms, as well as general psychopathology for people with schizophrenia within the past week. Symptom severity for each item is rated according to which anchoring points in the 7-point scale (1 = absent; 7 = extreme) best describe the presentation of the symptom. 7 Items, (minimum score = 7, maximum score = 49)

SECONDARY OUTCOMES:
Total Symptoms | 12 weeks
  Clinical Severity as determined by the Positive and Negative Syndrome Scale (PANSS) positive symptom subscale. The PANSS is a standardized, clinical interview that rates the presence and severity of positive and negative symptoms, as well as general psychopathology for people with schizophrenia within the past week. Symptom severity for each item is rated according to which anchoring points in the 7-point scale (1 = absent; 7 = extreme) best describe the presentation of the symptom. 30 Items, (minimum score = 7, maximum score = 210)
Negative Symptoms | 12 weeks
  Clinical Severity as determined by the Positive and Negative Syndrome Scale (PANSS) positive symptom subscale. The PANSS is a standardized, clinical interview that rates the presence and severity of positive and negative symptoms, as well as general psychopathology for people with schizophrenia within the past week. Symptom severity for each item is rated according to which anchoring points in the 7-point scale (1 = absent; 7 = extreme) best describe the presentation of the symptom. 7 Items, (minimum score = 7, maximum score = 49)
Cognition | 12 weeks
  As measured by the Penn Computerized Neurocognitive Battery (CNB)
Sheehan's disability scale (SDS) | 12 Weeks
  The SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life. Total score 0-30 (0 unimpaired, 30 highly impaired)
Global Assessment of Function (GAF) | 12 weeks
  The Global Assessment of Functioning, or GAF, scale is used to rate how serious a mental illness may be. It measures how much a person's symptoms affect his or her day-to-day life on a scale of 0 to 100.
Quality of Life Scale (QOL) | 12 weeks
  Self-administered questionnaire designed for use in patients with chronic illnesses. 7-point Likert-type scale ranging from "delighted" (7) to "terrible" (1). Total scale score (possible range: 16 - 112)

OTHER OUTCOMES:
Total Positive and Negative Syndrome Scale (PANSS) | 12 weeks
  Clinical Severity as determined by the Positive and Negative Syndrome Scale (PANSS) positive symptom subscale. The PANSS is a standardized, clinical interview that rates the presence and severity of positive and negative symptoms, as well as general psychopathology for people with schizophrenia within the past week. Symptom severity for each item is rated according to which anchoring points in the 7-point scale (1 = absent; 7 = extreme) best describe the presentation of the symptom. 30 Items, (minimum score = 7, maximum score = 210)
Penn Computerized Neurocognitive Battery (CNB) | 12 weeks
  Developed in the Brain Behavior Lab at Penn, the CNB is a series of computerized tests that measure accuracy and speed of performance in major domains of cognition, including social-cognition. Battery measures the executive functions of abstraction and mental flexibility, attention, and working memory, episodic memory for words, faces and figures, intellectual functioning including verbal and nonverbal reasoning and spatial orientation, facial emotion processing and sensorimotor and motor speed. The participant completes this test on the computer with oversight by a research team member.
Sheehan's disability scale (SDS) | 12 weeks
  The SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life. Total score 0-30 (0 unimpaired, 30 highly impaired)
Global Assessment of Function (GAF) | 12 weeks
  The Global Assessment of Functioning, or GAF, scale is used to rate how serious a mental illness may be. It measures how much a person's symptoms affect his or her day-to-day life on a scale of 0 to 100.
Quality of Life Scale (QOL) | 12 weeks
  Self-administered questionnaire designed for use in patients with chronic illnesses. 7-point Likert-type scale ranging from "delighted" (7) to "terrible" (1). Total scale score (possible range: 16 - 112)

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L. Nimgaonkar, M.D., Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No individual subject data will be shared.